CLINICAL TRIAL: NCT04680286
Title: The Use of Intraoperative Methadone in Children Undergoing Open Urological Surgery: a Randomized, Double-blind Trial
Brief Title: Intraoperative Methadone in Children Undergoing Surgery
Acronym: METACEBO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment due to covid-19 and organizational changes.
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23956082; 2020-002945-41 (EudraCT Number)
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-04

CONDITIONS: Pain, Acute; Pain, Postoperative; Children, Only
Keywords: methadone; analgesics; opioids; postoperative; placebo
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Methadone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomisation and study medication will be handled by the hospital pharmacy. All research team members, caregiving clinicians and enrolled patients will be blinded to the study allocation arms and the randomisation list will be concealed until all statistical analyses are made.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): A 5 ml syringe with saline will be prepared and study drug will be administered as intravenous bolus dose (0.1 mg/kg). The study drug will be administered at induction of anesthesia.
  Interventions: Other: Placebo
- Methadone (Experimental): A 5 ml syringe with 1 mg/ml of methadone will be prepared and study drug will be administered as intravenous bolus dose (0.1 mg/kg). The study drug will be administered at induction of anesthesia.
  Interventions: Drug: Methadone Hydrochloride

INTERVENTIONS:
Drug: Methadone Hydrochloride — Single dose, intravenous bolus, 0,1 mg/kg administered at induction of anesthesia.
  Other Names: Methadone
  Arms: Methadone
Other: Placebo — Single dose, intravenous bolus. Administered as the experimental arm.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
A prospective double-blind, randomized controlled trial investigating the effect of a single-dose of intraoperative methadone on postoperative pain and opioid consumption in 96 children undergoing open urological surgery.

DETAILED DESCRIPTION:
Treatment of postoperative pain is a challenge in younger children undergoing outpatient surgery. After discharge parents must assess pain intensity and administer analgesics, including opioids, as per needed. It has been shown that parents often hesitate to administer analgesics. The result is unrelieved pain that negatively affects the whole family and increases the risk of unscheduled contacts with healthcare professionals.

In children, methadone has shown a half-life of 19,2 +/-13,6 hours. Regarding outpatient surgery, methadone is an opioid with unique pharmalogical properties that may be advantageous. A single-dose of this long acting opioid administered perioperatively could provide a stable analgesia and potentially reduce the need for shorter-acting opioids in the PACU and at home.

ELIGIBILITY:
Inclusion Criteria:

Children scheduled for open urological surgery at the Outpatient Clinic at Aarhus University Hospital.

Exclusion Criteria:

* Age =/> 5 years at the date of operation
* Born preterm (Before gestational age of 37 weeks)
* Congenital heart disease
* Previous scrotal surgery
* Laparoscopic operation
* American Society of Anaesthesiologists (ASA) physical status lll, IV or V
* Allergy to study drugs
* Preoperative daily use of opioids
* Parents with inability to provide informed consent
* Severe respiratory insufficiency
* Acute abdominal pain
* Severe kidney insufficiency
* Treatment with rifampicin

Ages: 0 Years to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Patients consumption of analgesics in the PACU. | 3 hours
  Within the first 3 hours from extubation (or until discharge from PACU, if discharged before 3 hours).
Pain intensity (highest score) | 3 hours
  FLACC-score - Face, Legs, Activity, Cry og Consolability, 0-10, where 10 is the highest pain score. Within the first 3 hours from extubation (or until discharge from PACU, if discharged before 3 hours)

SECONDARY OUTCOMES:
Readiness to discharge | 6 hours
  Time for readiness to discharge from PACU assessed by PACU nurse.
Patients need of supplemental oxygen in PACU | 3 hours
  Need of supplemental oxygen within the first 3 hours after extubation,(or until discharge from PACU, if discharged before 3 hours)
Awakenings during the first night after discharge. | 24 hours
  Parents will answer whether the child have been awake and whether they believe the awakening(s) where due to pain.
Pain intensity the first postoperative day | 48 hours
  Assessed by parents, 3 FLACC-scores - Face, Legs, Activity, Cry og Consolability, 0-10, where 10 is the highest pain score, during the first postoperative day.
Analgesic consumption following discharge until evening on the first postoperative day | 36 hours
  From discharge until 8 PM the first day following surgery. Collected by parents.
Unscheduled parental contacts to the hospital | 4 days
  Parental contacts to hospital regarding pain and/or analgesics until 4 days following surgery.

OTHER OUTCOMES:
FLACC-scores - Face, Legs, Activity, Cry og Consolability, 0-10, where 10 is the highest pain score, at home | 48 hours
  Parental experience with assessment of the FLACC-score at home following discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT04680286/Prot_SAP_000.pdf